CLINICAL TRIAL: NCT03659435
Title: Open, Randomized, 2-period, 2-sequence, Cross-over Relative Bioavailability Study to Investigate the Pharmacokinetics and to Assess the Bioequivalence of a Rivastigmine Test Patch Formulation 9.5 mg/24 h (Twice Weekly Patch) Compared to the Reference Exelon® 9.5 mg/24 h (Once Daily Patch) Applied for 11 Days
Brief Title: Rivastigmine Bioequivalence Trial With Multiple Application of Transdermal Patches (9.5mg/24h)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1352riv18ct; 2018-001570-18 (EudraCT Number); C_30410_P1_05 (Other: Luye Pharma AG / Luye Supply AG)
Record Dates: First submitted 2018-08-28; First posted 2018-09-06 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RID-TDS 9.5 mg/24 h (Experimental): 3 consecutive applications of 1 patch (1st patch for 4 days, 2nd patch for 3 days, 3rd patch for 4 days) covering an 11-day period
  Interventions: Drug: RID-TDS 9.5 mg/24 h
- Exelon® 9.5 mg/24 h (Active Comparator): 11 consecutive applications of 1 patch (each patch will be applied for 1 day) covering an 11-day period
  Interventions: Drug: Exelon® 9.5 mg/24 h

INTERVENTIONS:
Drug: RID-TDS 9.5 mg/24 h — 3 consecutive applications of 1 patch (1st patch for 4 days, 2nd patch for 3 days, 3rd patch for 4 days) covering an 11-day period
  Arms: RID-TDS 9.5 mg/24 h
Drug: Exelon® 9.5 mg/24 h — 11 consecutive applications of 1 patch (each patch will be applied for 1 day) covering an 11-day period
  Arms: Exelon® 9.5 mg/24 h

SUMMARY:
The present clinical trial will be conducted in order to compare the bioavailability of rivastigmine and to assess bioequivalence at steady-state of the Test product RID-TDS 9.5 mg/24 h (Luye Pharma AG, Germany) and the marketed Reference product Exelon® 9.5 mg/24 h transdermales Pflaster (Novartis Pharma GmbH, Germany) after multiple patch application. Each of both treatments will last for 11 days with a washout period of 14 days between the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. sex: male
2. age: 18-55 years, inclusive
3. body-mass index2 (BMI): ≥18.5 kg/m² and ≤ 30.0 kg/m²
4. good state of health as determined by no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination (including vital sign) and/or ECG, as determined by the investigator
5. non-smoker or ex-smoker for at least 1 month
6. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient (especially sick sinus syndrome or conduction defects such as sino-atrial block, atrio-ventricular block)
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient (especially predisposition to urinary obstruction and seizures)
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient (especially active gastric or duodenal ulcers or predisposition to these conditions)
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. Subjects with chronic obstructive or other pulmonary diseases or bronchial asthma
6. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations or previous history of application site reactions suggestive of allergic contact dermatitis with rivastigmine patch
7. subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
8. systolic blood pressure < 90 or >139 mmHg
9. diastolic blood pressure < 60 or >89 mmHg
10. heart rate < 50 bpm or > 90 bpm
11. body weight below 50 kg
12. QTc interval > 450 ms
13. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
14. ASAT > 20% ULN, ALAT > 10% ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 μmol/l ULN).
15. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
16. Presence or history of acute or chronic diseases especially of the skin, which could affect dermal absorption or metabolism, which may interfere with the bioavailability and /or the pharmacokinetics of the IMP based on assessment of the investigator
17. Skin abnormality (e.g. tattoo or scar) at the application site
18. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
19. history of or current drug or alcohol dependence
20. positive alcohol or drug test at screening examination
21. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol per day
22. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
23. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
24. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
25. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
26. regular treatment with any systemically available medication
27. subjects practising top-performance sports (more than 4 x 2 h per week)
28. subjects suspected or known not to follow instructions
29. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
AUC96-264 | from 96 to 264 hours after the first patch application
  partial area under the plasma concentration vs. time profile for the time interval 96-264 hours
Cmax,96-264 | from 96 to 264 hours after the first patch application
  maximum concentration in plasma during the nominal time interval 96-264 hours
Cmin,96-264 | from 96 to 264 hours after the first patch application
  absolute minimum concentration within the nominal time interval 96-264 hours
Patch adhesion properties | at 96, 168 and 264 hours after the first Test patch application
  lower one-sided 90% confidence limit for the mean of Test

SECONDARY OUTCOMES:
Skin irritation | from first patch removal until last patch removal (approx. 9 to 13 days)
  frequency of scores for quantification of skin irritation per treatment and time point
Adverse events | approximately 7 to 12 weeks, through study completion in case of follow-up
  descriptive evaluation of frequency and intensity, relationship to the IMP, action taken, outcome, seriousness, period and treatment
inhibition of plasma butyrylcholinesterase (BuChE) | from first patch application until 24 hours after the last patch removal
  % inhibition of BuChE activity in plasma in comparison to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany